CLINICAL TRIAL: NCT04641949
Title: Methoxyflurane and Fentanyl in the Lower Body Negative Pressure Model of Hypovolemia in Healthy Volunteers; a Randomized, Placebo-controlled Crossover Study
Brief Title: Methoxyflurane and Fentanyl in LBNP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Lars Øivind Høiseth, Overlege, PhD, Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: lbnp_methoxy_fent_2019
Record Dates: First submitted 2020-11-18; First posted 2020-11-24 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Hypovolemia; Cardiac Output, Low; Analgesia
Keywords: Methoxyflurane; Fentanyl
MeSH Terms: conditions — Hypovolemia; Cardiac Output, Low; Agnosia | interventions — Lower Body Negative Pressure

STUDY DESIGN:
Intervention Model Description: Randomized, placebo controlled, crossover study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both drug interventions (intravenous fentanyl and inhaled methoxyflurane) will have NaCl placebo comparators. As the methoxyflurane has a characteristic smell, some drops of methoxyflurane will be placed on the exterior of the placebo methoxyflurane inhalation devices. Further, the subjects will rinse the mouth with a mouthwash shortly before inhalation to cover the taste of methoxyflurane.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Methoxyflurane (Active Comparator): Inhalation methoxyflurane 99,9%, 3 ml, single dose. Intravenous NaCl 9 mg/ml, XX ml, single dose.
  Interventions: Procedure: Lower body negative pressure (LBNP)
- Fentanyl (Active Comparator): Intravenous fentanyl 50 microgr/ml, XX ml, single dose Inhalation NaCl 9 mg/ml, 3 ml, single dose.
  Interventions: Procedure: Lower body negative pressure (LBNP)
- Placebo (Placebo Comparator): Intravenous NaCl 9 mg/ml, XX ml, single dose. Inhalation NaCl 9 mg/ml, 3 ml, single dose.
  Interventions: Procedure: Lower body negative pressure (LBNP)

INTERVENTIONS:
Procedure: Lower body negative pressure (LBNP) — LBNP is a model of experimental hypovolemia, whereby the lower body is exposed to negative pressure leading to sequestering of blood in the lower body and central hypovolemia. LBNP will be induced stepwise with increments of 10 mmHg, each level lasting 1 min. LBNP will be terminated at symptoms or signs of impending hemodynamic collapse.

SUMMARY:
The study is a single-centre, placebo-controlled, crossover study on healthy volunteers aiming to explore non-inferiority of methoxyflurane and fentanyl compared to placebo on the tolerance to hypovolemia.

DETAILED DESCRIPTION:
The study will explore the effects of fentanyl and methoxyflurane versus placebo (NaCl; saline) on the hemodynamic response to hypovolemia in healty volunteers. Hypovolemia will be induced in the "lower body negative pressure" model. XX healthy volunteers will be exposed to inhaled methoxyflurane, 3 ml or intravenous fentanyl, XX mg or placebo in a randomized order (cross-over) at least 3 days apart.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age.
* Must be below 65 years of age.
* Signed informed consent and expected cooperation for the study and follow up must be obtained and documented according to ICH GCP, and national/local regulations.

Exclusion Criteria:

* Any medical condition limiting physical excertional capacity or requiring regular medication (allergy and oral contraceptives excepted)
* Pregnancy
* History of syncope (syncope of presumed vasovagal nature with known precipitating factor excepted)
* Any known cardiac arrhythmia
* History of renal disease
* History of liver disease
* Previous substance abuse
* Allery or known serious side-effects to opioids or methoxyflurane

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Cardiac output | Measured continuously during LBNP-exposure.
  Cardiac output as measured by suprasternal Doppler and/ or non-invasive (volume clamp) pulse contour analysis.

SECONDARY OUTCOMES:
Time to hemodynamic decompensation | 15 minutes
  Time from start LBNP to symtomps or signs of hemodynamic decompensation (and termination of LBNP); defined by:
  * Symptoms of pre-syncope (light-headedness, nausea or sweating)
  * Mean arterial pressure-reduction to less than 75% of baseline for >3 s
  * Heart rate-reduction to less than 75% baseline for >3 s
Mean arterial pressure | Measured continuously during LBNP-exposure.
  Change in mean arterial blood pressure with increasing LBNP, as measured by the volume-clamp method.
Stroke volume | Measured continuously during LBNP-exposure.
  Change in cardiac stroke volume with increasing LBNP, as measured by suprasternal Doppler and/ or the volume-clamp method.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoiseth LO, Fjose LO, Hisdal J, Comelon M, Rosseland LA, Lenz H. Haemodynamic effects of methoxyflurane versus fentanyl and placebo in hypovolaemia: a randomised, double-blind crossover study in healthy volunteers. BJA Open. 2023 Jun 28;7:100204. doi: 10.1016/j.bjao.2023.100204. eCollection 2023 Sep. PMID 37638077